CLINICAL TRIAL: NCT06565910
Title: Bupivacaine Liposome Plus Bupivacaine or Ropivacaine for PENG Block on Post Operative Pain Management in Patients Undergoing Hip Arthroplasty: a Prospective, Randomized, Single Blind, Active Controlled Study
Brief Title: Bupivacaine Liposome Plus Bupivacaine or Ropivacaine for Pericapsular Nerve Group Block in Hip Arthroplasty (PENG)
Acronym: PENG
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Wei Mei, Clinical Professor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TJ-IRB202407066
Record Dates: First submitted 2024-08-09; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Femoral Neck Fractures; Femur Head Necrosis; Hip Fractures
Keywords: Bupivacaine Liposome; PENG block; Hip Arthroplasty; Randomized Controlled Trial
MeSH Terms: conditions — Femoral Neck Fractures; Femur Head Necrosis; Hip Fractures | interventions — Bupivacaine; Ropivacaine

STUDY DESIGN:
Intervention Model Description: This study utilizes a parallel interventional design, where participants undergoing hip arthroplasty surgery will be allocated into two separate groups. One group will receive liposomal bupivacaine plus bupivacaine as a regional anesthetic for Pericapsular Nerve Group (PENG) block, while the other group will receive ropivacaine for the same purpose. Both interventions will be administered under ultrasound guidance. The study aims to compare the analgesic efficacy, duration of pain relief, opioid consumption, and patient satisfaction between the two groups, with assessments conducted at multiple time points within 72 hours post-surgery. The parallel design allows for the direct comparison of the two interventions and their respective outcomes in managing postoperative pain following hip arthroplasty.
Who Masked: Participant, Outcomes Assessor
Masking Description: Given the distinct visual appearance of the liposomal bupivacaine (milky white) and ropivacaine (transparent), a double-blind study design is not feasible.
  Consequently, this study employs a single-blind approach where neither participants nor outcome assessors will be aware of treatment allocation. Healthcare providers administering the study drug will be aware of the treatment group assignment. Rigorous procedures will be implemented to minimize potential bias, including standardized outcome assessment tools, blinded data entry, and independent data analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liposomal Bupivacaine plus Bupivacaine Intervention (Experimental): Participants in this arm will receive liposomal bupivacaine(LB) plus bupivacaine(B) as a local anesthetic for PENG block under ultrasound guidance. Liposomal bupivacaine plus bupivacaine is being investigated for its analgesic effect in postoperative pain management following hip replacement surgery. This arm aims to evaluate the analgesic efficacy, duration of pain relief, and safety profile of liposomal bupivacaine plus bupivacaine compared to the standard local anesthetic, ropivacaine. Participants in this arm will undergo hip replacement surgery under spinal anesthesia and will be assessed for pain relief, opioid analgesic consumption, and any associated complications at multiple time points within 72 hours after surgery.
  Interventions: Drug: Liposomal bupivacaine plus bupivacaine
- Ropivacaine Intervention (Active Comparator): Participants in this arm will receive ropivacaine (R) as a local anesthetic for the PENG block under ultrasound guidance. Ropivacaine, a routinely used local anesthetic in clinical practice, is being compared to liposomal bupivacaine plus bupivacaine to assess its analgesic effect in postoperative pain management following hip replacement surgery. This arm aims to evaluate the analgesic efficacy, duration of pain relief, and safety profile of ropivacaine in comparison to the investigational intervention, liposomal bupivacaine. Participants in this arm will undergo hip replacement surgery under spinal anesthesia and will be assessed for pain relief, opioid analgesic consumption, and any associated complications at multiple time points within 72 hours after surgery.
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Liposomal bupivacaine plus bupivacaine — Liposomal bupivacaine is a prolonged-release formulation of the local anesthetic bupivacaine. This intervention involves the administration of liposomal bupivacaine plus bupivacaine as a local anesthetic for the pericapsular nerve group (PENG) block under ultrasound guidance. Liposomal bupivacaine is being investigated for its analgesic effect in postoperative pain management following hip replacement surgery. This formulation is designed to provide extended pain relief as compared to conventional bupivacaine formulations.
  Other Names: LB+B
  Arms: Liposomal Bupivacaine plus Bupivacaine Intervention
Drug: Ropivacaine — Ropivacaine is a commonly used local anesthetic in clinical practice, and it serves as the active comparator intervention in this study. Participants in the comparator arm will receive ropivacaine as a local anesthetic for the PENG block under ultrasound guidance.
  Other Names: R
  Arms: Ropivacaine Intervention

SUMMARY:
The goal of this clinical trial is to study the analgesic effect of liposomal bupivacaine plus bupivacaine for Pericapsular Nerve Group (PENG) block in postoperative pain management following hip replacement surgery. It will also assess the safety of liposomal bupivacaine for this purpose. The main questions it aims to answer are:

1. Is liposomal bupivacaine plus bupivacaine superior to ropivacaine in terms of analgesic efficacy, duration of pain relief, opioid consumption, and patient satisfaction?
2. What medical problems do participants encounter when using liposomal bupivacaine plus bupivacaine for PENG block in postoperative pain management following hip replacement surgery?

Researchers will compare liposomal bupivacaine plus bupivacaine to ropivacaine (a routinely used regional anesthetic in clinical practice) to determine if liposomal bupivacaine plus bupivacaine is more effective for pain management following hip replacement surgery.

Participants will:

1. Receive liposomal bupivacaine plus bupivacaine or ropivacaine as a regional anesthetic for PENG block under ultrasound guidance.
2. Undergo hip replacement surgery under spinal anesthesia.
3. Have pain relief, opioid analgesic consumption, and incidence of complications assessed at multiple time points within 72 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists(ASA) I~II
* Normal coagulation
* Clinical diagnosis of hip fracture

Exclusion Criteria:

* Presence of severe systemic diseases or ASA grade III or higher
* Allergy to amide local anesthetics

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Overall Opioid Consumption | this outcome will be monitored and recorded within 72 hours postoperatively
  This primary outcome entails tracking and assessing the total opioid consumption by participants following hip replacement surgery. The evaluation includes quantifying the amount of opioids prescribed and consumed by participants for pain management post-surgery. Opioid medications administered will be converted to morphine equivalents based on established conversion ratios. By analyzing overall opioid consumption, the study aims to evaluate the efficacy of the interventions in managing postoperative pain.

SECONDARY OUTCOMES:
Pain intensity | at multiple time points within 72 hours post-surgery.
  Pain intensity will be assessed using the Numerical Rating Scale (NRS), a 0-10 scale where 0 represents no pain and 10 represents the worst imaginable pain. Pain intensity will be measured at 10 time points: at baseline, 30min after PENG block, at Post Anesthesia Care Unit(PACU), 6 hours, 12 hours, and 24 hours 36 hours, 48 hours, 60 hours, 72 hours post-surgery.
Time to First Rescue Analgesic | 72 hours after surgery.
  Time to first rescue analgesic will be recorded as the interval from the end of the surgery to the administration of the first dose of rescue analgesic medication postoperatively.
Incidence of Complications or Adverse Events | 90 days after the surgical procedure
  This outcome focuses on monitoring and documenting any adverse events or complications that may arise as a result of the interventions, including liposomal bupivacaine and ropivacaine, during postoperative care following hip replacement surgery. The assessment involves the systematic identification, recording, and analysis of any untoward effects, adverse reactions, or complications experienced by participants attributable to the administered interventions. The aim is to evaluate the safety profile of both interventions and compare the incidence of complications between the treatment groups to ensure patient safety and well-being throughout the study period.
Duration of Hospital Stay | through study completion, an average of 1 year
  The duration of hospital stay is a significant secondary outcome that involves recording and comparing the length of time each participant remains hospitalized following hip replacement surgery. This outcome provides insight into the postoperative recovery process and the potential impact of the administered interventions, including liposomal bupivacaine and ropivacaine, on the participants' recovery trajectory. Assessing the duration of hospitalization allows for the evaluation of factors such as pain management, mobility, and postoperative care that may influence the participants' readiness for discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Mei, MD, Study Director — Department of Anesthesiology, Tongji Hospital, Tongji Medical College, HUST
Locations (1):
- Department of Anesthesiology, Tongji Hospital, Tongji Medical College, HUST, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
individual participant data sets to be shared will include all collected individual participant data that underlie the results reported in any publications resulting from the trial. This would typically include data related to pain relief, opioid analgesic consumption, incidence of complications, and any other relevant outcomes assessed at multiple time points within 72 hours after surgery.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: starting 6 months after publication.
Access Criteria: The IPD and any additional supporting information will be shared with qualified researchers upon request. Access will be granted for the purpose of conducting further analyses related to the outcomes of the clinical trial, such as but not limited to, pain relief, opioid analgesic consumption, and complications. Requests for access will be reviewed by the principal investigators and designated research personnel to ensure that the proposed analyses align with the objectives of the study and maintain participant confidentiality. Access to the data will be provided through a secure mechanism that safeguards the privacy and integrity of the individual participant data.

REFERENCES:
- [Background] Carmichael JC, Keller DS, Baldini G, Bordeianou L, Weiss E, Lee L, Boutros M, McClane J, Feldman LS, Steele SR. Clinical Practice Guidelines for Enhanced Recovery After Colon and Rectal Surgery From the American Society of Colon and Rectal Surgeons and Society of American Gastrointestinal and Endoscopic Surgeons. Dis Colon Rectum. 2017 Aug;60(8):761-784. doi: 10.1097/DCR.0000000000000883. No abstract available. PMID 28682962
- [Background] Temple-Oberle C, Shea-Budgell MA, Tan M, Semple JL, Schrag C, Barreto M, Blondeel P, Hamming J, Dayan J, Ljungqvist O; ERAS Society. Consensus Review of Optimal Perioperative Care in Breast Reconstruction: Enhanced Recovery after Surgery (ERAS) Society Recommendations. Plast Reconstr Surg. 2017 May;139(5):1056e-1071e. doi: 10.1097/PRS.0000000000003242. PMID 28445352
- [Background] Nelson G, Bakkum-Gamez J, Kalogera E, Glaser G, Altman A, Meyer LA, Taylor JS, Iniesta M, Lasala J, Mena G, Scott M, Gillis C, Elias K, Wijk L, Huang J, Nygren J, Ljungqvist O, Ramirez PT, Dowdy SC. Guidelines for perioperative care in gynecologic/oncology: Enhanced Recovery After Surgery (ERAS) Society recommendations-2019 update. Int J Gynecol Cancer. 2019 May;29(4):651-668. doi: 10.1136/ijgc-2019-000356. Epub 2019 Mar 15. PMID 30877144
- [Background] Batchelor TJP, Rasburn NJ, Abdelnour-Berchtold E, Brunelli A, Cerfolio RJ, Gonzalez M, Ljungqvist O, Petersen RH, Popescu WM, Slinger PD, Naidu B. Guidelines for enhanced recovery after lung surgery: recommendations of the Enhanced Recovery After Surgery (ERAS(R)) Society and the European Society of Thoracic Surgeons (ESTS). Eur J Cardiothorac Surg. 2019 Jan 1;55(1):91-115. doi: 10.1093/ejcts/ezy301. PMID 30304509
- [Background] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Background] McCann ME. Liposomal Bupivacaine. Anesthesiology. 2021 Feb 1;134(2):139-142. doi: 10.1097/ALN.0000000000003658. No abstract available. PMID 33433621
- See also: a description of liposomal bupivacaine: EXPAREL — https://www.exparelpro.com/?popup=false

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-09): https://cdn.clinicaltrials.gov/large-docs/10/NCT06565910/Prot_SAP_000.pdf
  • Informed Consent Form (2024-06-23): https://cdn.clinicaltrials.gov/large-docs/10/NCT06565910/ICF_001.pdf